CLINICAL TRIAL: NCT01644097
Title: A Phase II Feasibility and Correlative Study of Probiotic Supplementation in Cancer Patients Receiving Chemotherapy or Tyrosine Kinase Inhibitors (TKIs)
Brief Title: Probiotic Supplementation in Preventing Treatment-Related Diarrhea in Patients With Cancer Undergoing Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: issues with obtaining study product
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VAR0084; NCI-2012-01127 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Diarrhea; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Quality of Life
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (probiotic mix) (Experimental): Patients receive a mixture of Lactobacillus plantarum strain 299v, Bifidobacterium lactis probiotic supplement, and Lactobacillus acidophilus probiotic PO BID for 9 weeks. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: Lactobacillus plantarum strain 299v; Dietary Supplement: Lactobacillus acidophilus probiotic; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment; Dietary Supplement: Bifidobacterium lactis probiotic supplement
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID 9 weeks. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: placebo; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum strain 299v — Given PO
  Other Names: DSM 9843; Lp 299v
  Arms: Arm I (probiotic mix)
Dietary Supplement: Lactobacillus acidophilus probiotic — Given PO
  Arms: Arm I (probiotic mix)
Dietary Supplement: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Dietary Supplement: Bifidobacterium lactis probiotic supplement — Given PO
  Arms: Arm I (probiotic mix)

SUMMARY:
This randomized phase II clinical trial studies probiotic supplementation in preventing treatment-related diarrhea in patients with cancer undergoing chemotherapy. Probiotics may help prevent diarrhea caused by treatment with chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Incidence of moderate/severe (grade 2-4) diarrhea graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

II. Functional Assessment of Chronic Illness Therapy - Diarrhea (FACIT-D) Trial Outcome Index.

SECONDARY OBJECTIVES:

I. To evaluate the effects of probiotic supplementation on dose delays or reductions due to gastrointestinal (GI) toxicity.

II. To evaluate the effects of probiotic supplementation on anti-diarrheal medication use.

III. To evaluate the effects of probiotic supplementation on overall health-related quality of life (HR-QOL).

IV. To evaluate the effects of probiotic supplementation on febrile neutropenia.

V. To evaluate the effects of probiotic supplementation on adverse GI effects. VI. To evaluate the effects of probiotic supplementation on overall survival. VII. To evaluate the effects of probiotic supplementation on progression free survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive a mixture of Lactobacillus plantarum strain 299v, Bifidobacterium lactis probiotic supplement, and Lactobacillus acidophilus probiotic orally (PO) twice daily (BID) for 9 weeks. Treatment continues in the absence of unacceptable toxicity.

ARM II: Patients receive placebo PO BID 9 weeks. Treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a documented malignancy initiating treatment including (as a single agent or in combination with other drugs) any one of the following cancer therapeutics:

  o Fluorouracil (5FU), capecitabine, irinotecan, paclitaxel, docetaxel, cabazitaxel, crizotinib, sorafenib, sunitinib, erlotinib, or lapatinib
* Any pathologically confirmed malignancy for which the patient would receive any of the listed cancer therapeutics
* Performance status of Eastern Cooperative Oncology Group (ECOG) 0-2
* Patient must have an estimated life expectancy of at least 6 months
* Absolute neutrophil count (ANC) > 1500
* Platelets > 100K
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x ULN (upper limit normal)
* Serum bilirubin < 1.5 x ULN
* Serum creatinine < 1.5 x ULN
* Ability to understand and the willingness to sign a written informed consent document and comply with the treatment protocol

Exclusion Criteria:

* Patients currently undergoing treatment with the above listed therapeutics at time of initiation of trial; patients can have had prior treatment(s) with one or more of the agents if they are initiating a new treatment with another agent on the list, provided they have had at least a 2 week "washout" period
* Patients currently taking anti-diarrheal medications or therapy
* Patients undergoing hemodialysis
* Patients with known allergic or hypersensitivity reaction to probiotics, yoghurt, or similar diet or supplemental products
* Acute or chronic diarrhea, including lactose intolerance, gluten or other dietary sensitivity resulting in gastrointestinal symptoms
* Pregnant or nursing patients
* Known human immunodeficiency virus (HIV) positive
* Prior abdominal surgery resulting in a stoma, ostomy, fistula, or other anatomic defect
* Concurrent or near future radiotherapy; prior, completed radiotherapy allowed; any radiotherapy within the vicinity of the GI tract must have been completed at least 4 weeks prior to start of trial
* Treatment with any investigational drug within 4 weeks prior to enrollment
* Current treatment with antibiotics or other gut motility agents within 2 weeks of starting study medication
* Abnormal thyroid function that is not controlled with medication
* Patients taking other dietary supplements within 2 weeks of starting study medication
* Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2-4 diarrhea over the 9-week study period, assessed by CTCAE version 4.0 | Up to 9 weeks
  Will be calculated by the percentage of patients experiencing grade 2-4 diarrhea as documented by patient diary and primary oncologist's documentation. The data for patients on tyrosine kinase inhibitors and conventional cytotoxic chemotherapy will be analyzed both combined and separately.
FACIT-D Trial Outcome Index (TOI) | Up to 4 weeks post treatment
  The FACIT-D TOI has a range of scores from 0-100 which are a combination of physical well being, functional well being, and diarrhea subscale. The data for patients on tyrosine kinase inhibitors and conventional cytotoxic chemotherapy will be analyzed both combined and separately.

SECONDARY OUTCOMES:
Dose delays or reductions due to GI toxicity | Up to 9 weeks
Anti-diarrheal use | Up to 9 weeks
Overall HR-QOL | Up to 4 weeks post treatment
Febrile neutropenia | Up to 4 weeks post treatment
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 4 weeks post treatment
Overall survival | Up to 2 years
Progression free survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Russell Pachynski, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States